CLINICAL TRIAL: NCT06111625
Title: Short-term Blinatumomab as a Bridge Therapy for Hematopoietic Stem Cell Transplantation in B-cell Acute Lymphoblastic Leukemia With Low Leukemia Burden
Brief Title: Short-term Blinatumomab as a Bridge Therapy for Allo-HSCT in Low Burden B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Principle Investigator, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Blin-bridge 1.0
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Leukemia, Lymphoid
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blinatumomab (Experimental): Blinatumomab was administered via a peripherally inserted central catheter (PICC) with an initial dosage of 8 μg/day. The dosage gradually escalated to 28 μg/day, with a total dose of 175 μg, infused over 5 to 10 days. To mitigate the risk of cytokine release syndrome (CRS), dexamethasone at a dose of 20 mg was administered 12 hours before the onset of blinatumomab infusion. Patients underwent myeloablative conditioning therapy consisting of fludarabine-and-busulfan-based regimen. Peripheral stem cells from HLA-matched sibling donors (MSD), matched unrelated donors (MUD), or haploidentical donors (HID) were reinfused two days after conditioning. Follow-up examinations were scheduled at +1, +2, +3, +4, +6, +9, +12, +18, and +24 months post-transplant.
  Interventions: Drug: blinatumomab

INTERVENTIONS:
Drug: blinatumomab — Blinatumomab was administered via a peripherally inserted central catheter (PICC) with an initial dosage of 8 μg/day. The dosage gradually escalated to 28 μg/day, with a total dose of 175 μg, infused over 5 to 10 days. To mitigate the risk of cytokine release syndrome (CRS), dexamethasone at a dose of 20 mg was administered 12 hours before the onset of blinatumomab infusion.

SUMMARY:
The goal of this single-arm, prospective study is to test in low-burden B-cell lymphoblastic leukemia (B-ALL) patients undergoing allogeneic hemopoietic stem-cell transplantation (allo-HSCT). The main question it aims to answer is:

• The efficacy and safety of short-term blinatumomab as a bridging therapy to allo-HSCT in patients with low-burden B-ALL. Participants will take intravenous blinatumomab prior to allo-HSCT with an initial dosage of 8 μg/day. The dosage gradually escalated to 28 μg/day and continued for 5 to 10 days. Dexamethasone 20mg was administered 1 hour before the onset of blinatumomab infusion.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with B-ALL;
2. patients with age ≥ 16 years;
3. Availability of both pre- and post-transplantation disease status records.

Exclusion Criteria:

1. administration of blinatumomab therapy for more than 14 days;
2. patients with leukemia burden ≥ 10% before initiation of treatment;
3. patients with severe organ dysfunctions before treatment, including myocardial infarction, chronic heart failure, decompensated liver dysfunction, renal dysfunction, or gastrointestinal dysfunction;
4. patients with central nervous system leukemia.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Progression free survival of this group of patients at the end of 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival of this group of patients at the end of 2 years
Relapse rate | 2 years
  Relapse rate of this group of patients at the end of 2 years
Cumulative incidence of acute graft versus host disease (aGVHD) | Day +100
  Cumulative incidence of acute graft versus host disease (aGVHD) of this group of patients at day+100
Cumulative incidence of chronic graft versus host disease (cGVHD) | 2 years
  Cumulative incidence of chronic graft versus host disease (cGVHD) of this group of patients at the end of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No